CLINICAL TRIAL: NCT05035433
Title: A Prospective, Multicenter Clinical Study of the Effect of the Order of Dilatation of Papillary Muscle and Mechanical Lithotripsy on the Efficacy and Postoperative Complications of ERCP in the Treatment of Choledocholithiasis.
Brief Title: Effect of the Sequence of Dilatation and Lithotripsy on the Treatment of Choledocholithiasis With ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: RenJi Hospital (Other); Shanghai Pudong Hospital (Other)
Responsible Party: Principal Investigator, Xuefeng Wang, Chief surgeon of general surgery department, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XH-20-022
Record Dates: First submitted 2021-07-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Choledocholithiasis; Cholangiopancreatography, Endoscopic Retrograde
Keywords: Choledocholithiasis; Cholangiopancreatography, Endoscopic Retrograde; Lithotripsy; Endoscopic papillary balloon dilation
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First lithotripsy and then EPBD (Experimental): After successful selective bile duct intubation, contrast agent was injected to measure the thickness of the bile duct and the size of bile duct stones under fluoroscopy. For those meeting the inclusion criteria, sphincterotomy was performed first.Papillary sphincter incision after indwelling godet in bile duct, anti-popular character silk will be crushed stone on top into rubble after biliary tract, broken line to suitable size after the switch to expanding balloon EPBD and further kidney stones, papillary sphincter incision after indwelling godet in bile duct, anti-popular character silk will be crushed stone on top into rubble after biliary tract, broken balloon to suitable size after the switch to expansion, expansion size 10-12 mm, according to the lower bile duct diameter, expansion time of 30 seconds.Then, the stones were removed with a net basket or balloon, and the nasobiliary duct was placed to end the operation.
  Interventions: Procedure: First lithotripsy and then EPBD
- First EPBD and then lithotripsy (Experimental): After puncture of the papillary sphincter, the guide wire was indwelled in the bile duct, and the columnar dilating balloon was inserted in exchange. The dilation size was 10-12mm, and the dilation time was 30 seconds according to the diameter of the lower end of the bile duct.At the end of the expansion, the stones were broken to a suitable size using a one-piece gravel net basket.The calculi were removed by using a stone net basket or balloon, and the nasobiliary duct was placed to end the operation.
  Interventions: Procedure: First EPBD and then lithotripsy

INTERVENTIONS:
Procedure: First lithotripsy and then EPBD — After successful selective bile duct intubation, contrast agent was injected to measure the thickness of the bile duct and the size of bile duct stones under fluoroscopy. For those meeting the inclusion criteria, sphincterotomy was performed first.Papillary sphincter incision after indwelling godet in bile duct, anti-popular character silk will be crushed stone on top into rubble after biliary tract, broken line to suitable size after the switch to expanding balloon EPBD and further kidney stones, papillary sphincter incision after indwelling godet in bile duct, anti-popular character silk will be crushed stone on top into rubble after biliary tract, broken balloon to suitable size after the switch to expansion, expansion size 10-12 mm, according to the lower bile duct diameter, expansion time of 30 seconds.Then, the stones were removed with a net basket or balloon, and the nasobiliary duct was placed to end the operation.
  Arms: First lithotripsy and then EPBD
Procedure: First EPBD and then lithotripsy — After puncture of the papillary sphincter, the guide wire was indwelled in the bile duct, and the columnar dilating balloon was inserted in exchange. The dilation size was 10-12mm, and the dilation time was 30 seconds according to the diameter of the lower end of the bile duct.At the end of the expansion, the stones were broken to a suitable size using a one-piece gravel net basket.The calculi were removed by using a stone net basket or balloon, and the nasobiliary duct was placed to end the operation.
  Arms: First EPBD and then lithotripsy

SUMMARY:
Choledocholithiasis is a common and frequently occurring disease in China, accounting for 15.3% ~ 31.7% of the total cholelithiasis.According to its source, can be divided into primary and secondary choledocholithiasis.For large choledocholithiasis, it is difficult to remove all calculi after dilatation of large diameter balloon or mechanical stone following alone.Therefore, we used the method of balloon dilation combined with mechanical lithotripsy after EST.There are few researches on the sequence of balloon dilation and mechanical lithotripsy at home and abroad, and there is no unified standard.

Through the ERCP balloon expansion of duodenal papilla sphincter and mechanical lithotripsy in the treatment of common bile duct calculi in patients with clinical observation, the balloon expansion and mechanical lithotripsy time order of take stone, stone residues rate and the influence of recent complications such as postoperative pancreatitis, ERCP in the treatment of huge stones optimization procedure was formulated.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. For patients with choledocholithiasis found by MRCP and feasible ERCP lithotomy, the diameter of calculi ≥1cm should be indicated (number of calculi should be indicated >5 or<5)
3. During ERCP, the surgeon determined that the calculi should be removed by combining EPBD and mechanical lithotripsy, and the calculi could be removed by a single ERCP
4. Previous cholecystectomy or planned recent cholecystectomy or liver lobectomy can also be included
5. Subjects voluntarily participate in this study and sign the informed consent

Exclusion Criteria:

1. Coagulation disorders (INR>1.3) and peripheral blood plate count significantly decreased<50x10^9/L
2. Preoperative complicated with acute pancreatitis
3. Preoperative biliary hemorrhage
4. Complicated with severe liver disease and primary sclerosing cholangitis
5. Mirizzi syndrome and intrahepatic bile duct stones
6. Complicated malignant tumor of hepatobiliary and pancreatic system
7. Complicated with obvious stricture of the lower segment of the bile duct
8. intraoperative bile duct duodenal fistula was found
9. Previous EST or EPBD
10. Previous history of gastrointestinal reconstruction surgery 11. Other ERCP contraindications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-09-06 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Lithotomy time | About 20 minutes
  The time required from completion of papillary myotomy to completion of lithotomy, including the time of cylindrical balloon dilation
Stone residual rate | about 2 days
  Routine indwelling of the nasobiliary duct was performed, and nasobiliary angiography before removal was performed to confirm the presence of residual stones

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xuefeng, PhD, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China